CLINICAL TRIAL: NCT05320432
Title: Transcutaneous Electrical Nerve Stimulation for Pain Control During First Trimester Abortion: a Blinded Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation for Pain Control During First-trimester Abortion
Acronym: TENS 2 0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 62478
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Abortion in First Trimester; Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcutaneous electrical nerve stimulation (TENS) (Experimental): Prior to the procedure, the patient will have two sets of two self-adhesive electrodes placed parallel to the spinal cord at the T10-L1 and S2-S4 levels for TENS administration. For participants randomized to the experimental group, the non-blinded study coordinator will turn on the TENS unit 5 minutes prior to the procedure and monitor stimulating frequency level (80-100 Hz and pulse duration of 400 microseconds; intensity or frequency will be monitored to be administered to a non-painful level).
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Sham (Sham Comparator): For the participants randomized to sham, the same placement of electrodes will occur, but the unit will not be delivering electrical stimulation.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — A low-level electrical current through the skin activates the descending inhibitory systems in the central nervous system.
  Arms: Transcutaneous electrical nerve stimulation (TENS)
Device: Sham — No current applied through pads.
  Arms: Sham

SUMMARY:
First-trimester abortion aspiration procedures are painful and sedation is typically provided. It is unsafe to drive after sedation due to the prolonged motor delay from some anesthetic agents. Without a known escort, most clinics do not allow patients to use public transportation, taxis, or rideshare services. Arranging a ride may be harder for those seeking abortion care than other surgical procedures given privacy concerns and the need to travel far distances. Additionally, some people have medical reasons that makes sedation in an outpatient abortion clinic unsafe. As abortion restrictions increase and more people need to travel far distances to access care, it is important to investigate non-pharmacologic pain control options.

Transcutaneous electrical nerve stimulation (TENS) delivers a low-level electrical current through the skin. By activating the descending inhibitory systems in the central nervous system, these pulses of electrical current reduce sensitivity to pain. TENS has been shown to be effective in decreasing pain with menstrual cramps and during medication abortion, and it was found to be non-inferior to IV sedation for first-trimester procedural abortion. However, it remains unclear if TENS is better than ibuprofen and local anesthesia via paracervical block alone.

The overarching goal of this research is to identify an inexpensive, non-pharmacologic, alternative pain control strategy for those with a medical or social contraindication to IV sedation. The specific aim of this project is to evaluate the efficacy of TENS to prevent pain during first-trimester procedural abortion. To achieve this objective, a blinded, randomized superiority trial comparing the use of TENS to sham for management of pain during first-trimester aspiration abortion is proposed. This research is significant because the validation of a non-pharmacologic pain management technique would decrease barriers to accessing abortion care.

DETAILED DESCRIPTION:
Abortion is common: one in four individuals will seek this care during their reproductive lifetime. Most abortions occur in the first trimester and nearly all - greater than 95% - occur in the outpatient clinic setting. Uterine aspiration is painful; most patients desire additional analgesia beyond local anesthesia. However, not every patient is a candidate for office sedation since multiple medical conditions are a contraindication and patients must have a ride home. The prolonged motor delay from some anesthetic agents makes driving after sedation unsafe. Without a known escort to monitor for surgical and anesthetic complications as recommended by the American Society of Anesthesia, most clinics do not allow patients to use public transportation, taxis, or rideshare services. Arranging a ride may be harder for those seeking abortion care than other surgical procedures given privacy concerns and the need to travel far distances. As abortion restrictions increase and more people need to travel far distances to access care, it is important to investigate non-pharmacologic pain control options. Transcutaneous electrical nerve stimulation (TENS) delivers an electrical current through the skin to activate the descending inhibitory systems in the central nervous system, effectively reducing sensitivity to pain. A previous trial comparing TENS to IV sedation found similar postoperative pain scores with a significantly shorter recovery time in the TENS group; however, this study did not evaluate or report intraoperative pain scores. It was found in a randomized controlled trial comparing TENS to IV sedation (in conjunction with local anesthesia) for first-trimester surgical abortion and that TENS had non-inferior pain scores to IV sedation and was considered an acceptable modality for pain control among participants. Through this proposed double blinded randomized controlled trial, it is hoped to demonstrate that TENS is a superior, non-invasive alternative pain control option for people undergoing surgical abortion in the first trimester who otherwise are not eligible for or decline IV sedation. Ultimately, the hope is to identify an inexpensive, alternative, non-pharmacologic pain control strategy for those with a medical or social contraindication to IV sedation in an effort to decrease barriers to accessing abortion care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* English- or Spanish-fluency
* <12 weeks gestation
* Presenting for aspiration abortion

Exclusion Criteria:

* Planned use of oral or IV sedation
* Contraindications to office-based procedure as determined by attending physician
* Fetal demise
* Requiring pre-procedure use of misoprostol
* Contraindication to TENS units use (pacemaker or epilepsy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Started | 35 | 35
Completed | 35 | 33
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (6.5) | 29.9 (7.7) | 30.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 20 | 37
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70
Nulliparous [Count of Participants; unit: Participants] | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Pain During Cervical Dilation
Description: Pain with manual cervical dilation, assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intra-operative, collected during procedure (up to 30 seconds)
Population: Two excluded from sham as did not complete procedure.
Measure: Median (Full Range); unit: millimeters on VAS
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
millimeters on VAS | 44 [0 to 88] | 50 [0 to 96]

2. Secondary Outcome: Pain During Procedure
Description: Pain during aspiration assessed by visual analog scale (VAS, 0-100mm; 0 being "no pain" and 100 being "worst pain imaginable")
Time Frame: Intra-operative, collected during procedure (up to 30 seconds)
Population: Two participants excluded from sham - did not complete procedure
Measure: Median (Full Range); unit: millimeters on VAS
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
millimeters on VAS | 44 [0 to 100] | 56 [3 to 100]

3. Secondary Outcome: Overall Experience
Description: Patient experience assessed by visual analog scale (VAS, 0-100mm; 0 being "worst experience possible" and 100 being "best experience possible")
Time Frame: Post-operative, collected following procedure (up to 20 minutes)
Population: Two excluded from sham - did not complete procedure
Measure: Median (Full Range); unit: millimeters on VAS
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
millimeters on VAS | 75 [6 to 100] | 62 [0 to 100]

4. Secondary Outcome: Procedure Time
Time Frame: up to 20 minutes
Population: Two excluded from sham - did not complete procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
minutes | 7.3 (2.9) | 8.4 (4.1)

5. Secondary Outcome: Provider Perceived Ease of Procedure
Description: Provider experience assessed by visual analog scale (VAS, 0-100mm; 0 being "easiest to use" and 100 being "most difficult to use")
Time Frame: Post-operative, collected after procedure (up to 30 seconds)
Population: Two excluded from sham - did not complete procedure
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
score on a scale | 16 [2 to 62] | 15 [0 to 72]

6. Secondary Outcome: Time Spent in Recovery
Time Frame: up to 1 hour
Population: Two excluded from sham - did not complete procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
minutes | 25.4 (8.8) | 24.0 (10.8)

7. Secondary Outcome: Number of Participants Who Correctly Identified Whether They Received TENS or Sham
Description: This outcome is to measure the participant's perceived group allocation.
Time Frame: Post-operative, collected after procedure (up to 30 seconds)
Population: Two participants excluded from sham - did not complete procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
Number analyzed (Participants) | 35 | 33
Participants | 32 | 21

ADVERSE EVENTS:
Time Frame: 2 weeks post-procedure
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) | Sham
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT05320432/Prot_SAP_000.pdf